CLINICAL TRIAL: NCT06839781
Title: The Effect of Retirement Education According to Meleis' Transition Theory on Individuals' Retirement Planning and Quality of Life
Brief Title: The Effect of Retirement Education on Individuals' Retirement Planning and Quality of Life
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Principal Investigator, Sultan Kayan, Lecturer, Bilecik Seyh Edebali Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: BilecikSeyhEU-HEM-SK-01
Record Dates: First submitted 2025-02-07; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: quality of life; nursing; occupational health; transition theory

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not know whether they are in the intervention or control group. Data will be collected by an assistant researcher who is blind to the groups, statistical analyses will be performed by an independent statistician who is blind to the groups, and reporting will be completed without disclosing the coding used in the analysis. In this way, detection bias, statistical bias, and reporting bias will be controlled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Retirement Education Group (Experimental): This initiative is structured as a six-week training program designed to support individuals in adapting to the retirement process. By addressing various aspects of retirement, the program aims to ensure that participants transition into this phase of life in a well-prepared and informed manner. The first week will serve as an introduction, providing general information and initiating physical transition training. The second week will focus on health protection and development training. The third week will address social transition training. The fourth week will be dedicated to spiritual transition training. The fifth week will focus on financial transition training. The sixth and final week will bring together previously retired individuals and current participants. This program adopts a holistic approach, aiming to facilitate both the physical and psychosocial adaptation of individuals to the retirement process.
  Interventions: Other: Retirement education
- Control group (No Intervention): The control group is a group that will not receive any intervention on individuals who have similar characteristics to those in the intervention group. This group will receive 6 weeks of retirement training at the end of the study.

INTERVENTIONS:
Other: Retirement education — This initiative is structured as a six-week training program designed to support individuals in adapting to the retirement process. By addressing various aspects of retirement, the program aims to ensure that participants transition into this phase of life in a well-prepared and informed manner. The first week will serve as an introduction, providing general information and initiating physical transition training. The second week will focus on health protection and development training. The third week will address social transition training. The fourth week will be dedicated to spiritual transition training. The fifth week will focus on financial transition training. The sixth and final week will bring together previously retired individuals and current participants. This program adopts a holistic approach, aiming to facilitate both the physical and psychosocial adaptation of individuals to the retirement process.
  Arms: Retirement Education Group

SUMMARY:
The aim of this study is to learn the effects of retirement education applied to individuals aged 50 and over approaching retirement, according to Meleis's Transition Theory, on their retirement planning processes and quality of life.

The hypotheses of the study are as follows:

H01: There is no difference in retirement planning perception between the experimental group applied with Meleis's Transition Theory and the control group not applied in terms of retirement planning perception.

* There is no difference in financial planning perception of individuals in the experimental group applied with Meleis's Transition Theory and the control group not applied in terms of retirement education.
* There is no difference in psychosocial perception of individuals applied with Meleis's Transition Theory and retirement education in terms of retirement planning.
* There is no difference in health perception of individuals applied with Meleis's Transition Theory and retirement education in terms of retirement planning.
* There is no difference in lifestyle perception of individuals applied with Meleis's Transition Theory and retirement education in terms of retirement planning.

H02: There is no difference in quality of life between the experimental group applied with Meleis's Transition Theory and the control group not applied in terms of retirement education.

To evaluate the effectiveness of the training, researchers will collect data from the same number of people with similar characteristics at the beginning and end of the training.

Participants will (initiative group):

Answer the pre-test before the intervention Attend retirement education for 1 hour per week for 6 weeks Answer the post-test after the intervention Answer the follow-up test 1 month after the post-test

DETAILED DESCRIPTION:
Retirement refers to the end of working life after a long period of work, when there are difficulties in continuing the work done and a permanent income that means rewarding the labor is connected, and the rest of the life is spent without working. It represents an important life transition for the majority of older adults; the transition from a paid job to retirement is described as a complex, dynamic, longitudinal process. For this reason, individuals need to make retirement plans in order to facilitate adaptation to retirement. Many studies show that pre-retirement planning activities are associated with better physical and psychological health, higher life satisfaction, positive retirement attitudes, and adaptation to retirement. Retirement education refers to education provided to individuals on issues such as evaluating their free time and coping with the problems they will encounter during this period, with the aim of preparing them for retirement. Retirement education aims to help individuals develop positive attitudes about retirement; to easily adapt to this period physically, mentally, economically, and psychosocially; to continue their productivity during retirement, and to spend this period happily. In this context, retirement training to be provided will enable individuals who will retire to see the problems that come with retirement realistically; learn how to deal with these problems and minimize the negative effects of these problems. In order for the individual to embrace the idea of retirement and adapt to this period, retirement training should include consultancy services on issues such as physical, psychosocial, financial change and legal rights. Training on physical change should include topics such as aging and old age concepts, old age characteristics and problems (physical, psychological, cognitive, social), nutrition and diet, personal care, care for chronic diseases, protection and development of health. Training to be planned in the field of psychosocial change should include topics such as family support, role change and adaptation, time management, leisure activities, stress and coping methods, volunteer activities, civil society organizations, and the society's perception of the elderly. In financial change training, topics such as retirement salary and budget planning, additional income sources, re-employment opportunities, and management of health expenses should be addressed, while in training on legal rights, topics such as insurance and retirement severance pay, retirement investment funds and state contribution, and protection of personal data should be included. In the literature review, no nursing research was found that evaluated the effects of retirement education on retirement planning and health. In this context, our study has original value as it is the first study to address the retirement period, which is an important transition process, in the field of nursing.

This study aims to evaluate the impact of retirement education based on Meleis' Transition Theory on individuals approaching retirement. A randomized controlled experimental design following the CONSORT (Consolidated Standards of Reporting Trials) guidelines will be employed.

The research will be conducted in two factories located in the city center of Denizli. Both factories are institutionalized in the field of cable production and belong to the same employer. These institutions have been operating since 2006, primarily serving export markets. The factories were selected due to the predominance of employees aged 50 and above and the nature of the work, which involves heavy machinery operation. Factory A employs 514 individuals, while Factory B employs 471 individuals. The total number of administrative personnel in both factories is 19. The workforce is predominantly male, and work is conducted in shifts (07:00-15:00, 15:00-23:00, 23:00-07:00). Shift schedules are determined monthly, and employees rotate through all shifts. Both institutions have occupational health and safety specialists; however, regular health screenings and training activities are not conducted.

The study population consists of 247 individuals aged 50 and above working in both factories. The minimum sample size was determined using power analysis (G Power 3.1.9.4) with a power of 1-β=0.80, an alpha level of α=0.05, and an effect size of 0.26, resulting in 44 participants per group (44 in the intervention group and 44 in the control group), totaling 88 participants. To account for potential participant attrition, the minimum sample size was increased by 20%, bringing the final sample to 106 individuals (53 in the intervention group and 53 in the control group).

Inclusion criteria for the study are being literate, aged 50 and above, and having no communication impairments. Individuals who have previously received retirement education related to the study topics will be excluded. Termination criteria include missing two or more training sessions, becoming disabled during the study, or retiring.

A list containing information on the 247 employees aged 50 and above will be prepared. Participants will be assigned to experimental and control groups using a six-block combination method. Eighteen six-block combinations consisting of letters A and B will be generated by an independent researcher using the randomizer.org program. The 247 individuals will be assessed based on the inclusion and exclusion criteria, and eligible participants will be identified. The 106 participants required for the sample will be assigned to the intervention or control group according to the predetermined randomization blocks. Participants will not be informed of their group assignment. After an initial introduction meeting, participants' information will be collected, and they will be informed about the training process and the possibility of extended training duration to prevent them from discerning their group assignment. Data collection will be conducted by a research assistant unaware of the participants' group assignments. The researcher providing the training will meet the groups for the first time during the introduction meeting. Statistical analyses will be performed by an independent statistician blinded to the group assignments, and the analysis codes will remain undisclosed until the reporting is completed. This approach aims to control detection bias, statistical bias, and reporting bias.

Data will be collected using a Descriptive Information Form, the Retirement Planning Process Scale, and the World Health Organization Quality of Life Short Form (WHOQOL-BREF).

A training program will be developed covering the concept of retirement, changes occurring during retirement (physical, social, psychological), health protection activities and their benefits, and financial preparedness. Since no prior study in the field of nursing has focused on retirement preparation, six focus group interviews were conducted-three with six individuals planning retirement and three with six individuals who retired within the last five years. These interviews revealed a need and demand for education on physical, psychological, social, and financial aspects of retirement, guiding the development of the training content. The appropriateness, reliability, and quality of the training program will be evaluated by five experts. A pilot study with 10 individuals outside the study population will be conducted to assess the effectiveness of the training.

Due to the lack of similar studies on retirement education, relevant health protection and promotion studies were reviewed, revealing that training sessions typically range from 1 to 8 sessions with durations of 30-150 minutes. In this study, the retirement education will consist of six sessions, each lasting 60 minutes. To enhance effectiveness, training sessions will be conducted in groups of no more than 15 participants.

Before the intervention, a meeting will be held with the control group to explain the study's purpose. Baseline data will be collected using the Descriptive Information Form, the Retirement Planning Process Scale, and WHOQOL-BREF. After the intervention, post-test data will be collected, followed by follow-up test data one month later. Once follow-up data collection is completed, the control group will also receive retirement education, but no other interventions will be applied during the study period.

Following the control group, the intervention group will be introduced to the study. An introductory meeting will be held to provide information about the study's objectives and procedures. Baseline data will be collected using the Descriptive Information Form, the Retirement Planning Process Scale, and WHOQOL-BREF. The retirement education program will be conducted over six weeks, with one 60-minute session per week. Post-test data will be collected at the final session, followed by follow-up test data one month later.

The independent variable in this study is retirement education based on Meleis' Transition Theory, while the dependent variables include financial, lifestyle, psychosocial, and health perception levels related to retirement planning, as well as quality of life scores.

Data will be analyzed using IBM SPSS 26.0. The normality of continuous variables will be tested using the Kolmogorov-Smirnov test (n>50). The chi-square test will be used to compare dependent variables with independent variables. If parametric test assumptions (normality and homogeneity of variance) are met, numerical measurements between independent groups will be compared using the Independent Samples t-test; otherwise, the Mann-Whitney U test will be used. Descriptive statistics will be presented as mean ± standard deviation (x̄ ±SD) for parametric tests or as median and min-max values for non-parametric tests. Comparisons of two dependent groups will be performed using the Paired Samples t-test if parametric assumptions are met; otherwise, the Wilcoxon test will be applied. For categorical numerical data, comparisons of more than two dependent groups will be conducted using the Friedman test. A significance level of p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria for the Study

* Literacy
* Being over 50 years old
* Not having any verbal communication disabilities (language, speech, vision or -hearing problems) Retirement Planning Process Scale score falling outside the cut-off value Exclusion criteria for the study
* Having previously received retirement training on the subjects covered by the study Criteria for termination of the study
* Individual not attending two or more training sessions for any reason
* Individual retiring due to disability during the program period

Min Age: 50 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Pre-test (The Process of Retirement Planning Scale (PRePS)) | 1 months
  The scale consists of four sub-dimensions and 48 items, namely the financial planning process, lifestyle planning process, psychosocial planning process and health planning process, which evaluate the processes of planning for individuals to evaluate the increased free time during their retirement years, to ensure sufficient income, to maintain healthy social relations, to gain health protection and development behaviors, and to maintain positive relations with the family. The financial planning process sub-dimension consists of 14 items, the lifestyle planning process sub-dimension consists of 11 items, the psychosocial planning process sub-dimension consists of 12 items and the health planning process sub-dimension consists of 11 items. The scale is a five-point Likert type. Higher scores obtained from the scale indicate that the individual's frequency of retirement planning behavior increases.
Pre-test (World Health Organization Quality of Life Short Form (WHOQOL-BREF)) | 1 month
  It is a scale developed by WHO in 1998 to assess perceived quality of life. It consists of 4 sub-dimensions, namely physical, mental, social and environmental, and 26 items. In addition to 26 questions, the scale includes 1 national question (27th question). This question was evaluated within the environmental sub-dimension in the Turkish validity-reliability study. The scale includes 2 questions (1st-2nd questions) that assess quality of life and general health status, which are not included in the 4 sub-dimensions. The physical domain consists of 7 items, the psychological domain consists of 6 items, the social relationship domain consists of 3 items, and the environmental domain consists of 7 items. Each sub-dimension is scored on a Likert-type scale between 1-5, and there is no total score for the scale. Scores between 4-20 can be obtained from each sub-dimension.

CONTACTS AND LOCATIONS:
Locations (1):
- Bilecik Seyh Edebali University, Bilecik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No